CLINICAL TRIAL: NCT04234100
Title: Study of the Bioavailability of Hesperidine and Narirutin Provided by an Orange Juice to Identify Various Metabotypes in Prehypertensive and Hypertensive Grade 1 Individuals (FLAVOTIP)
Brief Title: Bioavailability of Hesperidine and Narirutin From Orange Juice to Identify Metabotypes in Hypertension
Acronym: FLAVOTIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technological Centre of Nutrition and Health, Spain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FLAVOTIP
Record Dates: First submitted 2020-01-13; First posted 2020-01-21 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Blood Pressure; Hypertension
Keywords: Hypertension; Flavonoids; Orange juice; Metabotypes
MeSH Terms: conditions — Hypertension | interventions — Hesperidin; narirutin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orange juice rich in hesperidin and narirutin (Experimental): The consumption of the orange juice will be made in a single dose of 500 ml. The juice is presented in a concentrated and frozen format, packed in opaque cans of 500 mL, for which it must be thawed and diluted with mineral water up to 1.5 L before its ingestion.
  Interventions: Other: Orange juice rich in hesperidin and narirutin

INTERVENTIONS:
Other: Orange juice rich in hesperidin and narirutin — The product is a concentrated orange juice provided by the CITRUS Department of Florida (USA: www.FloridaCitrus.org).

SUMMARY:
Flavonoids are polyphenolic compound mainly found in fruits and vegetables with numerous beneficial health effects as protection against cardiovascular diseases by an antihypertensive effect. The intestinal microbiota plays a key role in the metabolization of these compounds, so that differences in the composition and activity of the microbiota between individuals can generate different metabotypes. Flavonoids are found mainly in their conjugated form linked to the monosaccharide rhamnose and need to be metabolized by the intestinal bacteria, releasing the rhamnose, to be absorbed and, thus, bioactive. The bacterial enzyme responsible of rhamnose hydrolysis is α-L-rhamnosidase, whose activity can vary considerably depending on the composition of the microbiota. In fact, a great interindividual variability has been observed in the ability to absorb flavonoids, which allows to classify individuals according to the corresponding metabotype. In a previous project, the investigators confirmed the interindividual differences in the bioavailability of hesperidin and narirutin, two flavonoids naturally present in orange juice. However, the role of the intestinal microbiota in the metabolism of hesperidin and narirutin needs to be elucidated.

On this basis, the following hypothesis is presented: individuals with arterial hypertension can be classified into 3 different metabotypes that are the result of the ability to absorb hesperidin and narirutin, determined by the urinary excretion of their respective metabolites, and these metabotypes are associated with different microbiota enterotypes and with different fecal α-L-rhamnosidase activity.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women over 18 years of age
2. Systolic blood pressure ≤159 mm Hg
3. Sign the informed consent

Exclusion Criteria:

1. Body mass index (BMI) ≥ 35 kg / m2
2. Glucose > 126 mg / dL
3. Systolic blood pressure ≥ 160 mm Hg and diastolic blood pressure > 100 mm Hg or taking antihypertensive drugs
4. LDL cholesterol > 189 mg / dL
5. Triglycerides > 350 mg / dL
6. Anemia (hemoglobin ≤ 13 g / dL in men and ≤ 12 g / dL in women)
7. Tobacco addiction
8. Consumption of medicines, antioxidants or vitamin supplements 30 days before the study
9. Use of antibiotics during the last 30 days prior to the study
10. Consumption of prebiotics and / or probiotics during the 30 days prior to the study
11. Clinical history of gastrointestinal disease or presence of intestinal disorders at the time of inclusion
12. Chronic alcoholism
13. Monitoring a vegetarian diet
14. Pregnant or with intent to get pregnant
15. Being in breastfeeding period
16. Participation in a clinical trial or nutritional intervention study, in the last 30 days.
17. Inability to follow the study guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
Percentage of absorption of hesperidin and narirutin | After 24 hours of juice consumption
  Quantification of the metabolites derived from hesperidin and narirutin in basal and 24-hour urine samples, using Liquid Chromatography coupled to Mass Spectrometry (LC-QqQ).
  From the profile of metabolites detected in urine, the percentage of absorption of hesperidin and narirutin with respect to the amount ingested will be quantified to determine the metabotypes, based on the urinary excretion corresponding to each volunteer:

SECONDARY OUTCOMES:
Fecal α-L-rhamnosidase activity | Basal
  Quantification of α-L-rhamnosidase activity in fecal samples by incubation of the samples with the substrate p-nitrophenyl α-Lrhamnopyranoside and the subsequent measurement of the aborsbance to a length wavelength of 405 nM in a spectrophotometer.
Gut microbiota composition | Basal
  Metagenomic analysis in fecal samples. The bacteria DNA will be extracted and massive sequenced by the Ion Torrent platform.
  The relative abundances of the different bacterial populations will be determined in fecal samples at different taxonomic levels, and microbial diversity will be analyzed.
Enterotype classification | Basal
  Metagenomic analysis in fecal samples. The bacteria DNA will be extracted and massive sequenced by the Ion Torrent platform.
  Enterotypes will be analyzed to classify volunteers in 3 enterotypes based on their intestinal microbiota composition.
Creatinine levels | Basal and after 24 hours of juice consumption
  Quantification of creatinine concentration in basal urine and 24 hours urine samples by a colorimetric assay.

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Solà, Dr, Principal Investigator — UTNS(Eurecat_Reus)/HUSJR. Reus, Tarragona, Spain
Locations (1):
- Centro Tecnológico de Nutrición y Salud (Eurecat-Reus), Reus, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Technological Centre of Nutrition and Health. Eurecat_Reus — http://eurecat.org